CLINICAL TRIAL: NCT05167565
Title: Prospective Study to Investigate Changes in Both Brain and Behavior and Its Underlying Neural Correlates in Human Infants
Brief Title: Longitudinal Development of Behavior and Its Underlying Neural Correlates in Human Infants
Acronym: MultiLongDev
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL21_0921; 2021-A02238-33 (Other: ID-RCB)
Record Dates: First submitted 2021-11-25; First posted 2021-12-22 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Healthy Volunteers
Keywords: Beta burst activity; Cognitive and motor development; MRI; EEG; behavioral test; Diffusion tensor imaging (DTI); beta bursts
MeSH Terms: interventions — Diffusion Tensor Imaging; Glycation End Products, Advanced; Psychiatric Status Rating Scales

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Infants aged around 3 month (Experimental): 80 infants aged around 3 months will be included in this study up to around 12.5 months
  Interventions: Other: MRI/DTI; Other: EEG; Other: Eye Tracking; Other: Ages and Stages Questionnaire (ASQ); Other: Infant Behavior Questionnaire Revised (IBQ-R); Other: Beck Depression Inventory (BDI); Other: The Brief Fear of Negative Evaluation Scale (BFNE); Other: Edinburgh Postnatal Depression Scale

INTERVENTIONS:
Other: MRI/DTI — High resolution MRI scans will be acquired from each infant at three time points (~3, 6, and 12 months), while they are naturally asleep to measure the progressive myelination of the major brain fiber tracks, grey matter maturation, and to create generative models for source reconstruction of EEG sensor data.
Other: EEG — EEG will be used to record infant brain activity during reaching and grasping actions to analyze beta activity
Other: Eye Tracking — Infants will be presented with the experimental stimuli, which will consist of images of adults displaying different facial expressions and non-social images (e.g. a cross, a geometric pattern). This procedure is based on commonly used eye tracking paradigms designed to assess attention biases in infancy. Infant eye movement and position will be measured during stimuli presentation.
Other: Ages and Stages Questionnaire (ASQ) — The parents will be asked to complete the ASQ questionnaire (Developmental questionnaire).
  ASQ-3 has 5 aspects: Communication, Gross motor, Fine motor, Problem solving and Personal-Social Each aspect has 6 questions, if the answer is Yes, score = 10, Sometimes = 5 and Not yet = 0. ASQ-3 average = average score of 5 aspects.
Other: Infant Behavior Questionnaire Revised (IBQ-R) — The parents will be asked to complete the IBQ-R questionnaire (Developmental questionnaire).
  The 191-item instrument provides scores on 14 temperament scales which in turn cluster into 3 overarching factors: Positive Affectivity/Surgency, Negative Emotionality, and Orienting/Regulatory Capacity. Items are rated on a 7-point scale.
Other: Beck Depression Inventory (BDI) — The parents will be asked to complete the BDI questionnaire (Mental health questionnaire).
  Scale is a 21-item self-reported questionnaire which measures the existence and severity of symptoms of depression. Scores for each symptom are added up to obtain the total scores for all 21 items. Total score ranges from 0-63; of which 0-8 is considered no depression, 0-13 is minimal depression, 14-19 is mild depression, 20-28 is moderate depression and 29-63 is severe depression.
Other: The Brief Fear of Negative Evaluation Scale (BFNE) — The parents will be asked to complete the BFNE questionnaire (Mental health questionnaire).
  The BFNE measures anxiety associated with perceived negative evaluation. This scale is composed of 12 items describing fearful or worrying cognition. Scores from for each item are added up to obtain the total score.
Other: Edinburgh Postnatal Depression Scale — The parents will be asked to complete the Edinburgh Postnatal Depression Scale (Mental health questionnaire).
  This is a set of 10 screening questions that can indicate whether a parent has symptoms that are common in women with depression and anxiety during pregnancy and in the year following the birth of a child. The total score is calculated by adding the numbers selected for each of the 10 items. If the parent's score is 10 points or above, they should speak to a health professional about those symptoms.

SUMMARY:
The unique importance of human brain development during the first years of life is unquestionable. During an infant's first year, the brain undergoes its most dramatic structural and functional changes, with factors such as early social experience having a significant effect on this development. This study proposes to investigate changes in both brain and behavior across the first 12 months of life. At three time points (~3, 6, and 12 month), anatomical and diffusion magnetic resonance imaging (MRI), resting state functional magnetic resonance imaging (fMRI), electroencephalography (EEG), eye tracking, and observational data will be obtained from the same sample of infants. These measures will be used to track the development of important sensorimotor, socio-emotional, and cognitive skills and their underlying neural correlates, as well as investigate the effects of early social experience on specific aspects of this development

ELIGIBILITY:
Inclusion Criteria:

* Healthy newborns, boys and girls, aged 3 months
* Uncomplicated pregnancy and delivery, APGAR scores >8
* Full-term birth without identified neuromotor problems at birth
* No congenital or developmental anomalies affecting the brain
* No reported history of neurological disorders or learning disabilities in the infants
* No reported specific visual, developmental and cognitive impairment
* Absence of medication having a cerebral or psychological impact
* Both parents/ legal guardian must provide their consent and signature prior to participation of their infant in the study

Exclusion Criteria:

* Severe congenital malformation
* Infants requiring a corrective surgery
* Any refusal of a parent
* Infants with severe impairment of the general condition and vital functions
* Infants with dermatitis of the face or scalp
* Infants who receive neurological treatment
* Infants born pre-term (birth before 37 weeks gestation)
* Infants whose mothers have significant medical conditions and/or had significant complications during pregnancy
* Infants who are adopted,
* Infants who have a first degree relative with autism, intellectual disability, schizophrenia, or bipolar disorder,
* Infants who have any significant medical and/or genetic conditions affecting growth, development, or cognition,
* Infants who have any contraindication to MRI (metallic object, surgical material like cochlear implant)
* Maternal pre- eclampsia, placental abruption, maternal HIV status, and maternal alcohol or illicit drug use during pregnancy.

Min Age: 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-10-17 (Actual); Primary Completion 2026-01-28 (Actual); Study Completion 2026-01-28 (Actual)

PRIMARY OUTCOMES:
Fractional anisotropy | 9 months following the inclusion
  Integrity of white matter fiber tracts assessed by DTI measures of the mean fractional anisotropy (0-1, where 0=isotropic diffusion, 1=diffusion restricted along one dimension) along them.
Diffusivity | 9 months following the inclusion
  Integrity of white matter fiber tracts assessed by DTI measures of the mean, radial, and axial diffusivity (mm2/s) along them.
Regional myelination | 9 months following the inclusion
  Regional myelination assessed by T1 / T2 intensity ratios.

SECONDARY OUTCOMES:
Motor beta burst timing | 9 months following the inclusion
  The timing relative to movement onset (ms) of beta bursts in the motor cortex, measured with EEG.
Motor beta burst peak frequency | 9 months following the inclusion
  The peak frequency (Hz) of beta bursts in motor cortex, measured with EEG
Infant eye movement attentional bias | 9 months following the inclusion
  The proportion of time spent fixating to threatening (ABT) and positive (ABP) facial expressions relative to neutral, measured using eye-tracking.
Ages and Stages Questionnaire scores | 9 months following the inclusion
  Scores on the gross motor, fine motor, and personal-social aspects of the Ages and Stages Questionnaire (0-60, with higher scores indicating normal development).
Infant Behavioral Questionnaire Revised score | 9 months following the inclusion
  Scores on the approach, vocal reactivity, high intensity pleasure, smiling and laughter, activity level, perceptual sensitivity, sadness, distress to limitations, fear, falling reactivity / rate of recovery from distress, low intensity pleasure, cuddliness, duration and orienting, and soothability scales of the Infant Behavioral Questionnaire Revised (0-7, with high scores indicating higher levels on each temperament trait).
Brief Fear of Negative Evaluation total score | 9 months following the inclusion
  Total score on the Brief Fear of Negative Evaluation questionnaire (0-60, with higher scores indicating higher social anxiety)
Edinburgh Postnatal Depression Scale total score | 9 months following the inclusion
  Total score on the Edinburgh Postnatal Depression Scale questionnaire (0-30, with higher scores indicating more depressive symptoms)

CONTACTS AND LOCATIONS:
Locations (1):
- Institut des Sciences Cognitives (ISC) Laboratoire CNRS UMR6229, Bron, France